CLINICAL TRIAL: NCT03170297
Title: SC2i VIPER: EnVenomation Investigation Pilot to Evaluate Recovery
Acronym: VIPER
Status: Completed | Type: Observational
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency); Duke University (Other); Emory University (Other); Grady Health System (Other); Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: Pro00082061; HT9404-13-1-0032 (Other: HJF/USUHS)
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples collected will be used for quantification of over one hundred micro RNA (levels will be assessed) as well as multiple markers of inflammation such as Interleukins 1-36 and their receptors, interferons and their receptors, tumor necrosis factors and their receptors, CCL and CXCL family chemokines and their receptors, macrophage and granulocyte colony stimulating factors and their receptors, and lymphocyte secreted products related to the action of these proteins will be evaluated. No genetic testing will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Research interventions of blood sampling and data collection — Patient-Specific Functional Scale (PSFS) survey will be administered to patients to record symptoms at both the time of evaluation in the emergency department and in follow up by phone at 3, 7, 14, 21 and 28 days after discharge from the emergency department or hospital. The rest of the patients' care will be as usual care, and patients will have had research interventions of blood sampling and data collection as noted in the previously approved SC2i Tissue Data Acquisition Protocol (TDAP) Pro00054947 (ClinicalTrial.gov ID: NCT02182180).

SUMMARY:
The purpose of this study is to pilot data for a systematic molecular characterization of pathophysiologic perturbations incurred by snake envenomation and compare this to other inflammatory physiologic states such as trauma and sepsis. This sub-study will analyze samples of participants enrolled under the parent study "Surgical Critical Care Initiative Tissue and Data Acquisition Protocol".

DETAILED DESCRIPTION:
The goal of this study is to pilot data for a systematic molecular characterization of pathophysiologic perturbations incurred by snake envenomation and compare this to other inflammatory physiologic states such as trauma and sepsis. The investigators will characterize transcriptomic and immune biomarker response to varying clinical severities of snakebite envenomation and compare to that of sepsis and traumatic injury.

This sub-study will analyze samples of participants enrolled under a previously IRB-approved protocol, "Surgical Critical Care Initiative Tissue and Data Acquisition Protocol (SC2i TDAP)". All participants eligible for protocol SC2i TDAP (NCT 02182180) are eligible to be included in the current proposal, and conversely, the investigators will not enroll any participants in the current protocol who is not enrolled in SC2i TDAP. Participants enrolled under that protocol who have suffered snakebite envenomation will undergo additional procedure of follow up phone call 3, 7, 14, 21 and 28 days after discharge from the emergency department or hospital to fill out the PSFS via phone. All labs and other procedures will otherwise be as described in SC2i TDAP.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled into the Surgical Critical Care Initiative Tissue and Data Acquisition Protocol (NCT02182180) who have suffered a snakebite envenomation (enrolled under "Group 5: Non-traumatic conditions: individuals with non-traumatic causes of organ or system failure that mirror the phenotype of traumatic complications in Group 1") are eligible to be included in this study.
* Adult patients (18 years of age or older) in a manner that is sensitive to the inclusion of women and members of underserved minority groups.
* Potential participants or legally authorized representative (LAR) will be originally identified by clinical team, as described under Pro00054947 (NCT02182180). Only participants enrolled in Pro00054947 (NCT02182180) will be recruited for this sub-study

Exclusion Criteria:

* Pregnant women will be excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: -This study may analyze participants with snakebite envenomation along with similarly previously enrolled subjects who have suffered traumatic injury or sepsis who will serve as matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Survey and Data | 30 days after initial bite for the survey
  Patient Specific Functional Scale survey and piloting data for a systematic molecular characterization of pathophysiologic perturbations incurred by snake envenomation and compare this to other inflammatory physiologic states such as trauma and sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Elster, MD, Study Director — Uniformed Services University of the Health Sciences
Locations (1):
- Duke University Health Systems, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The PI will ensure that there is no unauthorized use of the data or samples. As this study is unblinded and nonrandomized it is felt that a formal Data Safety Monitoring Board is not necessary to insure the prompt implementation of patient safeguards. Data for this sub-study will be entered in a separate REDCap database, with data specific to this sub-study (i.e., PSFS, hospital re-admissions from phone follow-ups). This database will only be available to appropriately delegated key personnel. Any data shared outside of Duke key personnel will be de-identified,

REFERENCES:
- See also: Henry M. Jackson Foundation for the Advancement of Military Medicine — http://www.hjf.org
- See also: Uniformed Services University of Health Sciences — http://www.usuhs.edu
- See also: Duke University Medical Center — http://www.dukemedicine.org